CLINICAL TRIAL: NCT03853512
Title: Safety Assessment, Instrumental and Perceived Efficacy 21 Days of Use at Home - Bepantol Derma Spray® Dermal and Gynecological Acceptability Assessment.
Brief Title: A Study to Gain Information How Well Dexpanthenol Dermal Spray Helps the Skin to Recover After a Peeling in the External Genital Area of Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20507
Record Dates: First submitted 2019-02-15; First posted 2019-02-25 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Skin Recovery
Keywords: Dermal spray; Peeling; Skin hydration; Consumer satisfaction; Sensorial perception
MeSH Terms: conditions — Consumer Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women_Inguinal side BAY207543 (Experimental): Adult women apply BAY207543 to one side of the inguinal region, and semisolid vaseline to the the opposite side after skin peeling. The area with BAY207543 will be investigated.
  Interventions: Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray); Other: Semisolid vaseline
- Women_Inguinal side Vaseline (Active Comparator): Adult women apply BAY207543 to one side of the inguinal region, and semisolid vaseline to the the opposite side after skin peeling. The area with the vaseline will be investigated.
  Interventions: Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray); Other: Semisolid vaseline

INTERVENTIONS:
Drug: BAY207543 (Bepanthol, Bepantol® Derma Spray) — Product is applied to one side of the inguinal region.
Other: Semisolid vaseline — Product is applied to the other side of the inguinal region.

SUMMARY:
In this study, researchers want to learn more about the effect of dexpanthenol dermal spray on skin recovery after a dermatological procedure (peeling) in the intimate area of women.

After the peeling, participants will return within 3 weeks for 4 visits to the study center to investigate the skin conditions such redness, irritation, softness and possible side effects. In addition, study participants will be asked about their general acceptance of dexpanthenol dermal spray.

DETAILED DESCRIPTION:
The primary objective is to evaluate the efficacy of the test product to aid skin recovery after peeling in the female intima and inguinal region.

Secondary objectives comprise clinical efficacy with respect to skin hydration, softness, vitality, appearance etc. and skin recovery, consumer judgement of product performance and acceptability, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Phototypes I and II according to the Fitzpatrick scale;
* Participants willing to have peeling in the genital area to improve the general appearance of the skin and bleaching of spots.

Exclusion Criteria:

* Pathologies and/or skin injuries, such as psoriasis, sensitive skin, skin cancer, atopic dermatitis or other medical criteria to be considered at the time of evaluation
* Hyperpigmentation in the test area that interfere with the evaluation of possible reactions (vascular malformations, scars, increase of pilosity and large amount of nevi)
* Pathologies and/or active skin injuries (local and/or disseminated) in the evaluation area

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Transepidermal water loss by TEWL probe | Up to 23 days
  The transepidermal water loss (TEWL) is measured in g m2 h-1 with a Tewameter TM300.

SECONDARY OUTCOMES:
Skin properties of the participants | Up to 23 days
  Investigators assess various skin properties of the participants with a questionnaire (each scored from 1 to 5), resulting in an overall efficacy score from 12 to 60 (a higher score represents higher efficacy).
Treatment satisfaction | Up to 23 days
  Participants assess their treatment satisfaction with a questionnaire consisting of 19 items (each item is scored from 1-5) resulting in a score range of 19 to 95 (a higher score represents better treatment satisfaction).
Product evaluation | Up to 23 days
  Participants assess their sensorial perception of different product attributes (e.g. smell, absorption) with a questionnaire consisting of 6 items (each item is scored from 1-5) resulting in a score range from 6 to 30 (a higher score represents higher product satisfaction).
Number of adverse events by dermatological evaluation | Up to 23 days
Number of adverse events by gynecological evaluation | Up to 23 days
Severity of adverse events by dermatological evaluation | Up to 23 days
Severity of adverse events by gynecological evaluation | Up to 23 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medcin Instituto da Pele, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.